CLINICAL TRIAL: NCT01715142
Title: Evaluation of Tumoral Perfusion Modification by Dynamic Imaging After Chemotherapy Combining Gemcitabine and Nab-paclitaxel (Abraxane) in Patients With Potentially Operable, Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Effect on Tumor Perfusion of a Chemotherapy Combining Gemcitabine and Nab-paclitaxel (Abraxane) in Pancreatic Cancer
Acronym: NEOPAX-001
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jean-Luc Van Laethem (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Jean-Luc Van Laethem, MD, PhD, Erasme University Hospital
Organization: Erasme University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003592-19
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Adenocarcinoma Resectable; Pancreatic Adenocarcinoma Locally Advanced; Pancreatic Adenocarcinoma Metastatic
Keywords: Pancreatic cancer; Nab-paclitaxel; Gemcitabine; Neoadjuvant chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine+Abraxane (Experimental): Chemotherapy combining gemcitabine and Abraxane during 4 weeks (1 cycle) before surgery (cohort 1: resectable patients) and during at least 8 weeks (2 cycles or more in case of response of stable disease) (cohort 2: locally advanced and metastatic patients)
  Interventions: Drug: Gemcitabine; Drug: Abraxane

INTERVENTIONS:
Drug: Gemcitabine — Administrated intravenously at a dose of 1000 mg/m2 over 30 minutes weekly, on day 1, day 8, day 15 followed by one week of rest (before surgery of before starting of the next cycle depending on the cohort allocation)
  Other Names: GEMZAR
Drug: Abraxane — Administrated intravenously at a dose of 125 mg/m2 over 30 minutes weekly, on day 1, day 8, day 15 followed by one week of rest (before surgery of before starting of the next cycle depending on the cohort allocation)
  Other Names: nab-paclitaxel

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is a highly lethal disease with conventional treatments having little impact on disease course. Novel approaches are urgently needed to address inherent resistance to the current therapies and to identify new drugs or combinations that will have a high chance of success in pancreatic cancer patients. This proof-of-concept trial is studying the "dynamic" tumor response after the administration of a short course of gemcitabine and nab-paclitaxel (Abraxane) (a) during a window interval (4 weeks= 1 cycle) before surgery in resectable pancreatic cancer (cohort 1 = 21 patients) and (b) during at least 8 weeks (2 cycles) in locally advanced or metastatic pancreatic cancer (cohort 2 = 10 patients).

DETAILED DESCRIPTION:
Pancreatic cancer is a hypoperfused tumor, characterized by a high stroma density precluding cytotoxics delivery to the epithelial tumoral compartment. There is thus a rationale for combining chemotherapy and antistromal drugs like nab-paclitaxel (Abraxane), a solvent (Cremophor® EL)-free, albumin-bound form of paclitaxel that has been initially developed to reduce the toxicities associated with Taxol injection while maintaining or improving its chemotherapeutic effect. This unique protein formulation provides a novel approach of increasing intra-tumoral concentrations of the drug by a receptor-mediated transport process allowing transcytosis across the endothelial cell.

Abraxane has been approved for commercialization in 38 countries, including the US, Canada, the EU, Australia, China, India and Korea for the treatment of women with metastatic breast cancer. Abraxane alone and in combination is being evaluated in a number of cancers, including metastatic melanoma, non-small cell lung cancer, pancreatic cancer and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histo(cyto)logically proven ductal pancreatic adenocarcinoma;
* Resectable or potentially resectable tumor; resectability assessed during a multidisciplinary meeting with expert surgeon and radiologist (cohort 1), or locally advanced and/or metastatic tumor (cohort 2);
* First line chemotherapy;
* Age > 18 years;
* WHO performance status (PS) grade 0 or 1;
* Absolute neutrophil count > 1.5 x 10 9 / L, platelets > 100 x 10 9/ L, creatinine clearance (Cockcroft and Gault formula) > 60 ml/min, haemoglobin level > 10 g/dl (transfusions authorized), bilirubin<1.5 g/dl;
* Optimal biliary drainage;
* Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation of who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum or urine pregnancy test prior to treatment. All WCBP, all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study;
* Signed informed consent.

Exclusion Criteria:

* Previous anticancer therapy for the pancreatic adenocarcinoma;
* Biliary obstruction without endoscopic biliary drainage;
* Any contre-indication for surgery;
* Prior malignancy (except non-melanoma skin cancer, and in situ carcinoma of the uterine cervix treated with a curative intent and any other tumor in complete remission with a disease-free interval > 3 years);
* Uncontrolled congestive heart failure or angina pectoris, myocardial infarction within 1 year prior to study entry, uncontrolled hypertension (systolic pressure > 160 mm or diastolic pressure > 100 mm under well conducted antihypertensive treatment), QT prolongation;
* Major uncontrolled infection;
* Severe hepatic impairment;
* Any medical, psychological, or social condition, which, in the opinion of the investigator, could hamper patient's compliance to the study protocol and/or assessment/interpretation of the data;
* Pregnant or lactating women, or patients of both genders with procreative potential not using adequate contraceptive methods;
* Patients receiving or having received any investigational treatment within 4 weeks prior to study entry, or participating to another clinical study; patients previously enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03-21 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Dynamic tumor response rate as defined by a 40% modification of tumoral perfusion and cellular density parameters. | 4 weeks (duration of 1 cycle of neoadjuvant chemotherapy for resectable patients); 8 weeks (duration of 2 cycles of treatment for locally advanced and metastatic patients)
  In order to detect changes in the tumor microenvironment and to monitor treatment efficacy, Dynamic Contrast Enhanced-Magnetic Resonance Imaging (DCE-MRI) and Diffusion Weighted-Magnetic Resonance Imaging (DW-MRI) constitute tools more and more used. The acquired data can be analyzed using a pharmacokinetic model to obtain quantitative parameters relative to tissue perfusion and vascular permeability (Ktrans, a volume transfer constant of contrast agent between blood plasma and the extravascular extracellular space; Apparent Coefficient Diffusion as a surrogate marker of tissue cellularity). DCE/DW-MRI will be achieved before each chemotherapy treatment (and also before surgery for resectable patients). Each patient will be his/her own control by comparing serial imaging results with those of the baseline MRI.

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0. | 12 months
  Number of participants with (serious) adverse events will be considered as a measure of safety of the whole therapeutic sequence (gemcitabine+Abraxane+surgery for resectable patients; gemcitabine+Abraxane for locally advanced/metastatic patients)

OTHER OUTCOMES:
Tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria | 4 weeks (duration of 1 cycle of neoadjuvant chemotherapy for resectable patients); 8 weeks (duration of 2 cycles of treatment for locally advanced and metastatic patients)
Effect of treatment on selected biomarkers in tumor resection specimens (cohort 1) and in case of obtaining tissue by Endoscopic Ultrasound-Guided Fine Needle Aspiration (EUS-FNA) (cohort 2) | 4 weeks (duration of 1 cycle of neoadjuvant chemotherapy for resectable patients); 8 weeks (duration of 2 cycles of treatment for locally advanced and metastatic patients)
  Evaluation of biomarkers involved in gemcitabine and nab-paclitaxel activity : human equilibrative nucleoside transporter 1 (hENT1), deoxycytidine kinase (dCK), cytidine deaminase (CDA), secreted protein acidic and rich in cysteine (SPARC), taxanes-related biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Van Laethem, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (2):
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem, Antwerpen
  - Erasme University Hospital (ULB), Brussels